CLINICAL TRIAL: NCT02501694
Title: Enregistrement Des Bruits Vasculaires de l'artère Iliaque Externe Par STETHOscope électronique en Post - Effort Chez le SPORTif
Brief Title: Evaluation of Patients With Suspected Endofibrosis
Acronym: Stethosport
Status: Completed | Type: Observational
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2014-A00532-45
Record Dates: First submitted 2015-07-15; First posted 2015-07-17 (Estimated); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Peripheral Artery Disease
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Auditory Perception

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Auscultation — Electronic stethoscope

SUMMARY:
Define responses to exercise on both arterial bruits and oxymetry in patients referred for suspected endofibrosis.

DETAILED DESCRIPTION:
Recording of oxymetry during exercise and recovery. Recording of vascular bruits at rest ajnd post exercise.

ELIGIBILITY:
Inclusion Criteria:

Referred for exercise test -

Exclusion Criteria:

None

-

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Athletes referred for exercise tests
Sampling Method: Non-Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2018-10-01 (Actual)

PRIMARY OUTCOMES:
Caracteristics of sound | 1 day
  recording of sounds

CONTACTS AND LOCATIONS:
Overall Officials: Antoine BRUNEAU, MD, PhD, Principal Investigator — University Hopistal Angers, France
Locations (1):
- Centre hospitalier universitaire, Angers, France